CLINICAL TRIAL: NCT02522663
Title: The Impact of 24/7-phone Support on Readmission After Aortic Valve Replacement, a Randomized Clinical Trial
Acronym: AVRre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Bergesen Foundation (Other); Raagholt Foundation (Unknown); Norwegian Extra Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Stein Ove Danielsen, Research Fellow, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVRre
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Aortic Valve Disease
Keywords: telephone support; discharge management; readmission; aortic valve replacement
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Today, no post-discharge telephone support is offered as standard care from the hospital.
- Intervention group (Experimental): Experimental group is offered 24/7-telephone support during the first 1 month post-discharge, and patients are actively called at day 2 and day 9 day after discharge.
  Interventions: Other: 24/7-telephone support

INTERVENTIONS:
Other: 24/7-telephone support — ICU nurses answer the calls from treated AVR patients during the first month after discharge, and use an evidence-based information manual to answer questions from the patients.
  Arms: Intervention group

SUMMARY:
Aortic Valve Replacement (AVR) surgery for aortic valve disease continues to increase in numbers. With better surgical techniques and equipment, also older patients can be operated on, resulting in an growth of the older population. AVR is characterized by high rates of hospital readmissions, resulting in suboptimal care planning and higher health care costs. Hence, it is important to develop strategies to reduce hospital readmissions following AVR. The purpose if this study is to develop and test the efficacy of a 24/7-phone support in the reduction of readmissions after AVR treatment. Secondary outcomes are a reduced level of anxiety, less depressive symptoms and a better health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with AVR (biological or mechanical) single, AVR (b or m)+aortocoronary bypass, AVR (b or m)+supra coronary tube graft
* Can understand, speak and write native Language (norwegian), and be able to fill in the questionnaires
* Can be contacted by phone after discharge from hospital

Exclusion criteria:

* Patients who have been admitted to intensive care for more than 24 hours
* Patients who have complications related to surgery e.g. cerebral insult with significant impact on cognitive functions after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Reduced readmissions | 1 year follow-up
  Will use data from the national patient registry: Norway Patient Registry (NPR) and data from patient journals to measure the readmission rates. Main measure will be readmission rate 30 days after discharge for Aortic Valve Replacement (AVR).

SECONDARY OUTCOMES:
Reduced anxiety | 1 year follow-up
  Will use Hospital Anxiety and Depression Scale (HADS) for measuring outcome on anxiety. Measure times: T0: Before AVR, T1: 1 month after AVR, T2: 3 months after AVR, T4: 6 months after AVR, T5: 1 year after AVR
Reduced depression | 1 year follow-up
  Will use Hospital Anxiety and Depression Scale (HADS) for measuring outcome on depression. Measure times: T0: Before AVR, T1: 1 month after AVR, T2: 3 months after AVR, T4: 6 months after AVR, T5: 1 year after AVR.
Increased health related quality of life | 1 year follow-up
  Will use EQ-5D-3L questionnaire from The EuroQol Group to measure health related quality of life. Measure times: T0: Before AVR, T1: 1 month after AVR, T2: 3 months after AVR, T4: 6 months after AVR, T5: 1 year after AVR
Reduced costs | 1 year follow-up
  Will use data from the national patient registry: Norway Patient Registry, data from the patients journals and data from The Norwegian Health Economics Administration (HELFO). Cost-utility analysis to compare intervention group with the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Stein O Danielsen, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Danielsen SO, Moons P, Leegaard M, Solheim S, Tonnessen T, Lie I. Facilitators of and barriers to reducing thirty-day readmissions and improving patient-reported outcomes after surgical aortic valve replacement: a process evaluation of the AVRre trial. BMC Health Serv Res. 2020 Mar 27;20(1):256. doi: 10.1186/s12913-020-05125-5. PMID 32220252
- [Derived] Danielsen SO, Moons P, Sandvik L, Leegaard M, Solheim S, Tonnessen T, Lie I. Impact of telephone follow-up and 24/7 hotline on 30-day readmission rates following aortic valve replacement -A randomized controlled trial. Int J Cardiol. 2020 Feb 1;300:66-72. doi: 10.1016/j.ijcard.2019.07.087. Epub 2019 Jul 30. PMID 31387822
- [Derived] Lie I, Danielsen SO, Tonnessen T, Solheim S, Leegaard M, Sandvik L, Wisloff T, Vangen J, Rosstad TH, Moons P. Determining the impact of 24/7 phone support on hospital readmissions after aortic valve replacement surgery (the AVRre study): study protocol for a randomised controlled trial. Trials. 2017 May 30;18(1):246. doi: 10.1186/s13063-017-1971-y. PMID 28693599